CLINICAL TRIAL: NCT06672588
Title: Magnetic Seizure Therapy for Schizophrenia - Trial
Acronym: MAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2105
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Schizophrenia; Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Treatment Resistant Schizophrenia; Electroconvulsive Therapy; Magnetic Seizure Therapy; Convulsive Therapy
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double blind, parallel-group clinical trial with two treatment arms conducted at two academic institutions. The aim is to recruit 80 participants in the hope of having 50 participants complete the study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomized into the study using a permuted block method with a random number generator. The study statistician will prepare the randomization scheme. The block size will be fixed and study personnel will be blinded to the randomization block size.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic Seizure Therapy (MST) (Experimental): MST treatments will be administered using the MagPro MST with Cool TwinCoil.
  Interventions: Device: Magnetic Seizure Therapy (MST)
- Electroconvulsive Therapy (ECT) (Active Comparator): ECT treatments will be administered using the MECTA spECTrum 5000Q or MECTA Sigma.
  Interventions: Device: Electroconvulsive Therapy (ECT)

INTERVENTIONS:
Device: Magnetic Seizure Therapy (MST) — MST treatment will be administered using the MagPro MST with a Cool TwinCoil over the frontal cortex in the midline position using 100 Hz stimulation at 100% machine output. Seizure threshold will follow prior protocols used for frontal MST. Patients will receive care and be managed by anaesthesia as per standard ECT practice.
  Other Names: MST
  Arms: Magnetic Seizure Therapy (MST)
Device: Electroconvulsive Therapy (ECT) — In the ECT arm treatment, the MECTA spectrum 5000Q or MECTA sigma machine will be used. The ECT determination of seizure threshold and the adjustment of energy at subsequent sessions will be based on a standard published protocol. All participants will receive RUL-UB ECT at six times the seizure threshold. Patients will receive care and be managed by anaesthesia as per standard ECT practice.
  Other Names: ECT
  Arms: Electroconvulsive Therapy (ECT)

SUMMARY:
This trial aims to assess the clinical effects and tolerability of Magnetic Seizure Therapy (MST) as an alternative to electroconvulsive therapy (ECT) for Treatment Resistant Schizophrenia (RS).

DETAILED DESCRIPTION:
The study will involve a randomized, double blind, non-inferiority clinical trial with two treatment arms conducted in two academic institutions (the Centre for Addiction and Mental Health (CAMH) in Toronto, and University of British Columbia (UBC) Hospital in Vancouver, British Columbia). The investigators will compare MST to right unilateral ultrabrief pulse ECT (RUL-UB-ECT). Treatment will be administered two to three days per week. Clinical response will be assessed with the 18-item Brief Psychiatric Rating Scale (BPRS). Response will be defined as greater than or equal to 40% decrease in the BPRS positive psychotic symptom subscale (4 items - hallucinatory, behavior, suspiciousness, conceptual disorganization, and unusual thought content). Patients who do not meet response criteria after 15 treatment sessions will be considered non-responders and will cease treatment sessions. The blind will not be broken to participants until the completion of the entire study.

ELIGIBILITY:
Inclusion Criteria:

1. are inpatients or outpatients;
2. demonstrate capacity to consent according to the MacArthur competence assessment tool for clinical research (MacCAT-CR);
3. have a DSM-5 diagnosis of Schizophrenia or Schizoaffective Disorder for at least 2 years, as determined by the MINI International Neuropsychiatric Interview - Version 7 (MINI-7.0);
4. are 18 years of age or older;
5. have demonstrated resistance to at least 2 antipsychotics of 600 mg of chlorpromazine equivalents for at least 6 weeks;
6. have a BPRS score at baseline of at least moderate severity (>4) on one of the four psychotic items (i.e., hallucinatory behavior, suspiciousness, conceptual disorganization, unusual thought content) or at least 12 on these 4 items combined;
7. are considered to be appropriate to receive convulsive therapy as assessed by an ECT attending psychiatrist and a consultant anaesthesiologist;
8. are on an antipsychotic at an adequate dose and are agreeable to keeping their current antipsychotic treatment constant during the acute phase of the intervention;
9. are able to adhere to the intervention schedule;
10. meet the MST safety criteria;
11. If a woman of child-bearing potential: is willing to provide a negative pregnancy test and agrees not to become pregnant during trial participation.

Exclusion Criteria:

1. have a history of MINI diagnosis of a substance use disorder (other than nicotine and caffeine) within the past three months;
2. have a concomitant major unstable medical illness;
3. are pregnant or intend to get pregnant during the study;
4. have probable dementia based on study investigator assessment;
5. have any significant neurological disorder or condition likely to be associated with increased intracranial pressure or a space occupying brain lesion, e.g., cerebral aneurysm;
6. present with a serious medical condition,
7. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
8. require a benzodiazepine with a dose > lorazepam 2 mg/day or equivalent or any anticonvulsant due to the potential of these medications to limit the efficacy of both MST and ECT;
9. are unable to communicate in English fluently enough to complete the neuropsychological tests;
10. have a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) Response (18-Version) | Greater than 8 treatments (2.5 weeks)
  The scale is used to quantify psychiatric symptoms such as anxiety, depression, hallucinations, and unusual behaviours. The scale range is 18-126. A lower score indicates lower severity in anxiety, depression, and positive psychotic symptoms. A higher score indicates higher severity in negative and positive psychotic symptoms.
MATRICS™ Consensus Cognitive Battery (MCCB) | Greater than 8 treatments (2.5 weeks)
  The MCCB Assessments: The battery of cognitive assessments (ten in total) is intended to provide evaluation of key cognitive domains relevant to schizophrenia and related disorders and be a measure of cognitive change before and after the treatment course. The ten tasks focus on the following cognitive domains: speed of processing; attention/vigilance; working memory; verbal learning; visual learning; reasoning and problem solving; and social cognition.

SECONDARY OUTCOMES:
Scale for Suicidal Ideation (SSI) | Greater than 8 treatments (2.5 weeks)
  This scale is used to assess the presence or absence of suicidal ideation and the degree of severity of suicidal ideas. The scale range is 0 - 38 (total score). Lower scores indicate lower severity of suicidal ideation (i.e., better outcome). Higher scores indicate higher severity of suicidal ideation (i.e., worse outcome).
The Calgary Depression Scale for Schizophrenia (CDSS) | Greater than 8 treatments (2.5 weeks)
  CDSS is a nine item clinician rated outcome measure that assesses the level of depression in people with schizophrenia. It distinguishes depressive symptoms from negative positive and extrapyramidal symptoms. The scale range is 0 - 27. A lower score indicates lower severity in depressive symptoms. A higher score indicates higher severity in depressive symptoms.
Autobiographical Memory Test (AMT) | Greater than 8 treatments (2.5 weeks)
  Interviewer-rated measure with 10 items that indexes autobiographical memory recall and specificity.
Montreal Cognitive Assessment (MoCA) | Greater than 8 treatments (2.5 weeks)
  The MoCA is a 30-point screening test that takes approximately 10 minutes to administer. It assesses executive functioning, visuospatial abilities, memory, attention, working memory, language, and orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, M.D., MSc., Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - University of British Columbia Hospital, Vancouver, British Columbia
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this project will be used for future research by internal and external project collaborators. Deidentified participant data along with data dictionaries will be made available and to gain access data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months and ending 3 years after publication of the primary outcome paper.

REFERENCES:
- See also: Information About Research At the Centre for Addiction and Mental Health — https://www.camh.ca/en/science-and-research